CLINICAL TRIAL: NCT07255092
Title: Pain and Itch Neuromodulation: Effects of Offset Analgesia, Placebo, and Nocebo and Topographical Distribution of Itch and Pain Receptors
Brief Title: Mechanisms Underlying the Nocibo Effect of Contagious Itch. in Both Histaminergic and Nonhistaminergic Itch
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Associate Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20250017 Project 3
Record Dates: First submitted 2025-11-20; First posted 2025-11-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: ITCH
MeSH Terms: interventions — Histamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contagious itch (Experimental): A contagious itch will be induced by a video (without audio) showing people scratching.
  Interventions: Other: Histamine; Other: Cowhage (Mucuna Pruriens); Other: Placebo

INTERVENTIONS:
Other: Histamine — To deliver histamine, standard allergy skin prick test (SPT) lancets are applied
Other: Cowhage (Mucuna Pruriens) — The spicules will be manually inserted. Approximately 30-35 spicules are gently rubbed into a 1 cm diameter skin area on the forearm/face
Other: Placebo — To deliver steril water, standard allergy skin prick test (SPT) lancets are applied

SUMMARY:
The study consists of one experimental session of approximately 1½ hours. The participant will fill in a series of questionnaires about how you perceive itch and pain, and about some traits of your personality, such as depression, anxiety and stress. Afterwards, three areas will be selected on each forearm of the subjects.

Two areas will be treated with histamine, two with cowhage, and two with vehicle. One application of each substance will be conducted including the contagious itch component. During the 10 minutes of the application of the pruritogens, itch and pain will be continuously monitored using a VAS scale.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other drugs
* Previous or current history of neurological, immunological, musculoskeletal, cardiac disorder or psychiatric diagnoses that may affect the results (e.g., neuropathy, muscular pain in the upper extremities, anxiety, depression, schizophrenia, etc.)
* Moles, wounds, scars, or tattoos in the area to be treated or tested
* Current use of medications that may affect the trial such as antihistamines and pain killers
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain and itch
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical studies)
* Contraindications to capsaicin, including intolerance to chili or burns or wounds at the application site
* The subject is assessed as unable to engage in the necessary cooperation required by the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Measuring pain by computerized Visual Analog Scale Scoring | Immediately after the intervention
  The investigators will ask the subjects to rate the sensation of pain on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates" no pain" and 100 indicates "worst pain imaginable".
Measuring itch by computerized Visual Analog Scale Scoring | Immediately after the intervention
  The investigators will ask the subjects to rate the sensation of itch on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no itch" and 100 indicates "worst itch imaginable".

SECONDARY OUTCOMES:
Pain Catastrophizing Scale (PCS). | Baseline
  The PCS assesses negative and exaggerated coping concerning anticipated or experienced painful stimuli. Thirteen items have to be answered on a 5-point Likert-type scale ranging from 0 (Not at all) to 4 (all the time).
Itch Catastrophizing Scale (ICS) | Baseline
  The ICS assesses negative and exaggerated coping concerning anticipated or experienced itchy stimuli. Thirteen items have to be answered on a 5-point Likert-type scale ranging from 0 (Not at all) to 4 (all the time).
Learned Helplessness Scale (LHS) | Baseline
  The questionnaire consists of 20 items, and the participant's response to each item is rated on a 4-point Likert scale ranging from strongly agree (1) to strongly disagree (4).
Depression, Anxiety, Stress Scale (DASS-21) | Baseline
  The questionnaire measures the magnitude of depression, anxiety, and stress. Each of these three subscales consists of 7 questions answered using a 0-3 Likert scale, with 0 meaning "it did not apply to me", and 3 meaning "it applied to me very much"
Reinforcement Sensitivity Theory - Personality Questionnaire (RST-PQ). | Baseline
  The RST-PQ contains in total 65 items must be answered on a 4-point Likert (Strongly disagree → Strongly agree)
Positive And Negative Affect Schedule (PANAS) | Baseline
  Twenty words are associated with the subject's current feelings and have to be rated on a 5-points Likert-type scale from very slightly or not at all to extremely
Difficulties in Emotion Regulation Scale Short Form (DERS-SF) | Baseline
  The questionnaire is an 18-item measure used to identify emotional regulation issues in adults. Participants rate each item on a 5-point Likert scale (from 1 to 5) from almost never to almost always
Emotion Regulation Questionnaire (ERQ) | Baseline
  This questionnaire is designed to assess individual differences in the habitual use of two emotion regulation strategies: cognitive reappraisal and expressive suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree), where 4 means (neutral).

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Gistrup, Denmark, Denmark